CLINICAL TRIAL: NCT04271969
Title: Clinical Effectiveness Of High Frequency Chest Wall Oscillation (HFCWO) In A Bronchiectasis Population
Acronym: HFCWO
Status: Completed | Type: Observational
Sponsor: Electromed, Inc. (Industry)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: HFCWO-001
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Bronchiectasis
Keywords: HFCWO; Bronchiectasis; SmartVest
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: SmartVest Airway Clearance System — Pulmonary airway clearance of retained mucus via high frequency chest wall oscillation (SmartVest)

SUMMARY:
The primary objective is to compare the patient's baseline QoL prior to HFCWO use against the patient's QoL at various study timepoints over a one-year period of HFCWO use.

DETAILED DESCRIPTION:
This study will use a prospective interventional comparative study design using the patient's quality of life (QoL) as the primary study endpoint to determine HFCWO affect. The study will compare the patient's QoL baseline (established at enrollment prior to HFCWO treatment) to the QoL measured at various timepoints (enrollment, 2 months, 6 months and 12 months) over a one-year period whilst receiving HFCWO treatment. In addition, a baseline for the secondary endpoints will established at enrollment for comparison to measurements taken at various timepoints over a one-year period whilst receiving HFCWO treatment. The patient's medical records will be used to establish prior histories of exacerbation rates for comparison to exacerbation rates experienced after one year of HFCWO treatment. Patients will serve as their own control.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Previous diagnosis of bronchiectasis confirmed by HRCT within the last 6 months
3. Patients must have at least 6 months of medical records related to bronchiectasis
4. Patients must be stable and currently on a standard of care regimen for bronchiectasis such as hypertonic saline and/or PEP
5. Patients with 1 or more exacerbations within the last 12 months
6. Previous and existing productive cough
7. No previous HFCWO use

Exclusion Criteria:

1. Patients who are known to have cystic fibrosis
2. Patients who are known to have primary ciliary dyskinesia (PCD)
3. Patients with chronic obstructive pulmonary disease (COPD) without bronchiectasis
4. Patients breathing via an artificial airway
5. Severe bronchospasm based on exam or history
6. Any comorbidity(ies) or contraindications that would normally complicate tolerating HFCWO treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL): Quality of Life-Bronchiectasis (QOL-B) questionnaire | 1 year
  The primary endpoint is the subject's quality of life (QoL) using the Quality of Life-Bronchiectasis (QOL-B) questionnaire as the measurement tool. QoL measured at enrollment (baseline) will be compared to QoL measured at 2 months, 6 months and 1 year.
  The previously validated questionnaire is titled "Quality of Life Questionnaire - Bronchiectasis". The Likert style questionnaire asks the subject to subjectively rank their symptoms using a 4 scale base ranging from "a lot of difficulty" to "no difficulty" and "always" to "never".

SECONDARY OUTCOMES:
Clinical Measurements | 1 year
  1. Exacerbation rates
     a. Pre HFCWO exacerbation rates will be established by review of the patient's medical records. Post HFCWO will recorded at 2 months, 6 months and 1 year.
  2. Exacerbation frequency
     1. The time to the subject's next exacerbation will be recorded for comparison pre to post HFCWO
     2. Lung function (FEV1, FVC, FEF25-75) measured by standard spirometry
     3. Sputum production measured by using the Breathlessness, Cough and Sputum Scale (BCSS) questionnaire
     4. Patient adherence to HFCWO treatment measured by SmartVest Connect wireless feature
     5. Six-minute walk test measured using American Thoracic Society standard test guidelines/protocol
     6. Radiographic changes compare patient's original high-resolution computerized tomography (HRCT) taken to initially

CONTACTS AND LOCATIONS:
Overall Officials: George Solomon, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama - Birmingham (UAB University Hospital), Birmingham, Alabama
  - Emory University School of Medicine, Atlanta, Georgia
  - Temple University, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No